CLINICAL TRIAL: NCT07310251
Title: Effect of Conventional Warm-up Regarding to Stretching Warm-up on Physical Performance in Children Soccer Players
Brief Title: Conventional Warm-up on Physical Performance in Children Soccer Players
Acronym: RCT
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica del Maule (Other)
Responsible Party: Principal Investigator, Pablo Valdés-Badilla, PhD. in Physical activities science, Universidad Católica del Maule
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 23136643/2023
Record Dates: First submitted 2025-12-01; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Children Soccer Players
Keywords: Child; soccer; sports; players

STUDY DESIGN:
Intervention Model Description: This randomized crossover trial will investigate the acute effects of four different warm-up protocols on physical performance in male child soccer players
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Conventional warm-up condition (Experimental): The CC performed a traditional soccer warm-up for 10 minutes, consisting of 4 minutes of jogging in different directions at moderate to vigorous intensities, measured using the 10-point perceived exertion scale (RPE) scale, starting between 3 and 5 points and ending between 6 and 8 points, followed by movements performed in matches (jumps, ball kicks, changes of direction) distributed in three sets of 60 seconds each with a 60-second rest between sets. This condition did not include flexibility exercises.
  Interventions: Other: conventional warm-up regarding to stretching warm-up
- Static stretching condition (Experimental): The SSC consisted of a warm-up with static stretching for 10 minutes. Four stretching exercises were performed, one for each lower body muscle group (quadriceps, glutes, hamstrings, and triceps sural), distributed in two sets of 30 seconds each with a 45-second rest per exercise, performing progressive increases in joint range of motion. The intensity started between 3 and 5 points, ending between 6 and 8 points on the RPE scale
  Interventions: Other: conventional warm-up regarding to stretching warm-up
- Dynamic stretching condition (Experimental): The DSC consisted of a 10-min warm-up with dynamic stretching. Four stretching exercises were performed, one for each lower body muscle group (quadriceps, gluteus, hamstrings and triceps surae) distributed in two series of 30 s each with a rest of 45 s per exercise, dynamically executing oscillatory stretching movements with progressive increases in speed. The intensity started between 3 and 5 points, ending between 6 and 8 points of RPE.
  Interventions: Other: conventional warm-up regarding to stretching warm-up
- Ballistic stretching condition (Experimental): The BSC consisted of a warm-up with ballistic stretching for 10 min. Four stretching exercises were performed, one for each muscle group of the lower body (quadriceps, gluteus, hamstrings and triceps surae) distributed in two series of 30 s each with a rest of 45 s per exercise in which an elongated position was maintained for 5 s then 5 s of oscillation with progressive increments until completing the 30 s of each series. The intensity started between 3 and 5 points, ending between 6 and 8 points of RPE.
  Interventions: Other: conventional warm-up regarding to stretching warm-up

INTERVENTIONS:
Other: conventional warm-up regarding to stretching warm-up — The warm-up protocol was based on the guidelines of a previous study conducted on adolescent players in Chile. The CC performed a traditional soccer warm-up for 10 minutes, consisting of 4 minutes of jogging in different directions at moderate to vigorous intensities, measured using the 10-point perceived exertion scale (RPE) scale, starting between 3 and 5 points and ending between 6 and 8 points, followed by movements performed in matches (jumps, ball kicks, changes of direction) distributed in three sets of 60 seconds each with a 60-second rest between sets. This condition did not include flexibility exercises.
  The SSC consisted of a warm-up with static stretching for 10 minutes. Four stretching exercises were performed, one for each lower body muscle group (quadriceps, glutes, hamstrings, and triceps surae), distributed in two sets of 30 seconds each with a 45-second rest per exercise, performing progressive increases in joint range of
  Other Names: usual care

SUMMARY:
Considering the importance of an optimal warm-up to enhance performance in key soccer-related variables such as jump height, sprint speed, and ball kicking velocity, most available evidence to date has focused on youth and adult players, with limited studies conducted in children. Therefore, this study aimed to assess and compare the effects of a conventional warm-up and warm-ups including static stretching condition (SSC), dynamic stretching condition (DSC), and ball-specific condition (BSC) on jump performance countermovement jump (CMJ), squat jump (SJ), and drop jump (DJ) as well as on curve sprint speed, the Illinois change of direction test (ICODT), and ball kicking speed in male child soccer players. We hypothesized that the dynamic stretching warm-up would produce superior performance across most variables compared with the other conditions, due to its potential benefits for neuromuscular activation and optimization of the stretch shortening cycle.

DETAILED DESCRIPTION:
This randomized crossover trial will investigate the acute effects of four different warm-up protocols on the physical performance of youth soccer players. Participants will complete four warm-up conditions in random order: (i) conventional warm-up (CC), without flexibility exercises; (ii) static stretching condition (ESE); (iii) dynamic stretching condition (EDD); and (iv) ballistic stretching condition (ESC). Each condition will be separated by a 72-hour rest period.

After each warm-up, participants will undergo jump performance assessments including countermovement jump (CMJ), squat jump (SJ), and drop jump (DJ), corner sprint speed, agility using the Illinois Change of Direction Test (ICODT), and striking velocity with their dominant and non-dominant legs. Anthropometric measurements (height, body mass, and BMI) will be obtained according to ISAK standards. Warm-up protocols will be standardized to 10 minutes and their intensity will be adjusted using the Rate of Perceived Exertion (RPE) scale, progressing from moderate intensity (3-5 points) to vigorous intensity (6-8 points). Data normality will be verified using the Shapiro-Wilk test, and differences between conditions will be analyzed using a one-way ANOVA with Bonferroni post hoc correction. Effect sizes will be calculated using Cohen's d, with statistical significance at p < 0.05.

This study will aim to determine which warm-up method most effectively improves key soccer performance variables (jumping ability, sprinting, agility, and striking speed) in children, providing evidence for optimizing pre-competition routines in youth soccer.

ELIGIBILITY:
Inclusion Criteria:

* Male children aged 8 - 13 years, enrolled in a soccer school affiliated with amateur clubs in Chile.
* Regular participation in organized soccer training (≥2 sessions per week) for at least six months prior to the study.
* Absence of musculoskeletal or neurological injuries that could limit the ability to perform the warm-up or physical performance assessments.
* Availability of appropriate sports clothing and footwear for testing sessions.
* No concurrent participation in other soccer schools or competitive teams during the study period.
* No official matches or competitions scheduled on the same days as the experimental sessions.
* Signed assent and informed consent provided by the participant and a parent or legal guardian, respectively.

Exclusion Criteria:

* Sustain an injury or illness during the study period that prevents participation in testing.
* Fail to complete all four experimental conditions or physical assessments.
* Demonstrate non-compliance with the warm-up instructions or assessment procedures.

Ages: 8 Years to 13 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 20 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2026-05-18 (Estimated); Study Completion 2026-08-20 (Estimated)

PRIMARY OUTCOMES:
Bipedal height | 8 Weeks
  Bipedal height was measured using the Frankfort plane in a horizontal position, with a tape measure (Bodymeter 206, SECA, Germany; accuracy to 0.1 cm) attached to the wall
Body mass | 8 weeks
  Body mass was measured using an electronic scale (Omron HBF 514, Osaka, Japón; accuracy to 0.1 kg), while BMI was calculated by dividing body mass by bipedal height squared (kg/m2).
Jump performance | 8 weeks
  All jump tests were performed according to previous recommendations. For the CMJ, soccer players performed maximum effort jumps on an Ergojump® Globus mobile contact platform (ErgoTest, Codogne, Italy) with their arms resting on their iliac crests. Takeoff and landing were standardized at the exact location, and players performed full knee and ankle extensions during the flight phase. For the SJ, players stepped onto the contact platform with their arms on the iliac crest and knees semi-flexed at a 90° angle and the "stop" signal; the player maintained this posterior position, performing the maximum jump. Takeoff and landing were standardized at the exact location, and players performed full knee and ankle extensions during the flight phase. In the DJ test, participants were instructed to minimize ground contact time (<250 ms) after stepping off a 20 cm box. The best of three jumps (with a 1-
Curve sprint speed | 8 weeks
  Sprint time was assessed to the nearest 0.01s using single-beam timing gates Brower® Timing System, (Salt Lake City, Utah, United States of America). The test consisted of placing a "semicircle" at a distance of 17 m outside the large area of the soccer field, which is standardized as follows: a radius of 9.15 m from the penalty spot, a distance of 14.6 m from the starting point to the end in a straight line, an angle of 105.84° measured from the penalty spot, and a total distance of 17 m (determined by trigonometric analysis). Photocells were installed at both ends of the semicircle to determine the time it took the players to run the curve. The test started from the left side, and the participant had to run at maximum speed until crossing the finish line. Two attempts were evaluated in both directions of the curve (left and right), recording the results as "dominant side" and "non-dominant side," depending on the dominance of the children soccer player's lower
Agility | 8 weeks
  The dimensions and route markings for the Illinois Change of Direction Test (ICODT) were adjusted to established methods. The ICODT consists of placing four markers to indicate an area of 10 m by 5 m. In the center of the area, four markers are placed at 3.3 m from each other. The children soccer players start in a prone position with their chin touching the surface of the starting line. They accelerate for 10 m, turn around, return to the starting line, zigzag in and out of the four markers, and finally complete a second 10 m sprint to finish the ICODT speed test. Players were instructed to run around the markers rather than cross them. If a participant did not follow these instructions, the test was terminated and restarted after a 3-minute recovery period. Performance results were collected using Brower® Timing System single-beam timing gates (Salt Lake City, Utah, United States of America).
Ball kicking speed | 8 weeks
  Participants performed a maximal instep ball strike with their dominant and non-dominant legs after a two-stride run using a size five soccer ball (Molten Vantaggio 5000®, FIFA PRO certified, Hiroshima). Maximum speed was measured with a radar gun Speed (Gun SR3600, Sports Radar®, Homosassa, Florida, United States of America). Three attempts were carried out, recording the best of the three with a 1-min rest between each attempt. The data obtained for ball kicking speed was determined to have high reliability of 0.92.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica del Maule, Talca, Talca, Chile

IPD SHARING:
Plan to Share IPD: Undecided